CLINICAL TRIAL: NCT01624987
Title: Intervention to Support the Reintegration of Former Combatants and Soldiers
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Konstanz (Other)
Collaborators: World Bank (Other)
Responsible Party: Principal Investigator, Susanne Schaal, Susanne Schaal, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WB_2012
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Appetitive Aggression; Post-traumatic Stress Disorder
Keywords: Treatment of ex-combatants; FORNET for ex-combatants; Appetitive Aggression; Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- NET for Forensic Offender Rehabilitation (Experimental): Narrative Exposure Therapy for Forensic Offender Rehabilitation (FORNET)
  Interventions: Behavioral: NET for Forensic Offender Rehabilitation (FORNET): a variant of Narrative Exposure Therapy; Other: Control group

INTERVENTIONS:
Behavioral: NET for Forensic Offender Rehabilitation (FORNET): a variant of Narrative Exposure Therapy — During the proposed therapy, the client constructs a chronological narrative of his or her whole life which includes all traumatic experiences and perpetrated violent acts. All emotions, cognitions, sensory information, and physiological reactions are activated and linked to the autobiographical context.In five sessions the trained therapist and the client try to go through all important traumatic experiences and perpetrated violent acts. The sixth session is a group session with four to five clients. The group session is oriented on Interpersonal Psychotherapy and focuses on the role change from soldier to civilian.
Other: Control group — The control group receives no intervention.

SUMMARY:
The project aims to investigate if trauma-related disorders and appetitive aggression can be reduced in former ex-combatants in DR Congo when a specific intervention (Narrative Exposure Therapy for Forensic Offender Rehabilitation, FORNET) is delivered by trained local personnel (phase 1). In a second step, the project aims to investigates the treatment success if this specific therapy is carried out by local personnel who have been trained by other local personnel ("train the trainer", phase 2) under the supervision of experts of the University of Konstanz.

DETAILED DESCRIPTION:
The reintegration of former child soldiers and ex-combatants is a big challenge in war-torn countries. Former child soldiers and ex-combatants often suffer from mental health problems and show enhanced levels of aggression. The present study focuses on the reduction of appetitive aggression and the improvement of mental health in former child soldiers and ex-combatants in DR Congo.

The project consists of four steps:

1. Training of selected DDRRR personnel(first generation)in FORNET (a variant of Narrative Exposure Therapy to treat trauma-related disorders and to reduce appetitive aggression)by experts from the University of Konstanz.
2. Treatment phase 1: Intervention will be carried out by therapists of the first generation. The trained therapists of the first generation will be supervised from the experts of the University of Konstanz.
3. Training of a second generation of DDRRR personnel in FORNET by the therapists of the first generation.
4. Treatment phase 2: Intervention will be carried out by therapists of the second generation. The trained therapists of the second generation will be supervised from the therapists of the first generation.

The study is conceived as a randomized controlled study. In phase 1 and in phase 2, study participants will be randomized allocated to the intervention group (FORNET) and the control group (no intervention). The treatment effect will be measured by pre-post and 6-months follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Ex-combatants who live in a transit camp in Goma, Congo.

Exclusion Criteria:

Ages: 16 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Appetitive Aggression (Appetitive Aggression Scale) | 6 months
Symptoms of post-traumatic stress disorder (Post-traumatic Diagnostic Scale, PDS) | 6 months

SECONDARY OUTCOMES:
Symptoms of depression (Patient Health Questionnaire (PHQ-9) | 6 months
Functionality (Work and Social Adjustment Scale) | 6 months
Substance abuse | 6 months
Re-integration questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Elbert, Prof. Dr., Study Director — University of Konstanz
Locations (1):
- Transit Camp for ex-combatants/Reintegration camp for ex-combatants (ETN), Goma, Republic of the Congo